CLINICAL TRIAL: NCT01386723
Title: End of EXTEND: Observing for Sustained Response Despite Discontinuation of Medication in Patients With Persistent and Chronic Immune Thrombocytopenia (ITP) Treated With Eltrombopag
Brief Title: End of EXTEND: Discontinuation of Medication for Patients With Immune Thrombocytopenia
Status: Terminated | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 1003010950
Record Dates: First submitted 2011-06-13; First posted 2011-07-01 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Immune Thrombocytopenia
Keywords: eltrombopag; promacta; immune thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Discontinuation of eltrombopag: ITP subjects who have discontinued the use of eltrombopag
  Interventions: Drug: Discontinuation of eltrombopag

INTERVENTIONS:
Drug: Discontinuation of eltrombopag — Observation of subjects as they discontinue the use of eltrombopag
  Other Names: eltrombopag, promacta

SUMMARY:
This study proposes to observe whether a stable platelet count would be maintained without additional treatment in the long term in at least a proportion of patients who have discontinued eltrombopag taken for at least 4 months. This requires that if patients stop treatment with eltrombopag, they are not immediately transitioned to further treatment unless it is necessary.

The objective of the study is to assess how frequently patients who have discontinued eltrombopag attain a stable, treatment-free, unmaintained adequate platelet count 4 to 8 weeks after discontinuing eltrombopag and how long such a response lasts (if it occurs).

ELIGIBILITY:
Inclusion Criteria:

* A subject is eligible for study entry if all of the following criteria apply:

  * Subject or their guardian has signed and dated a written informed consent
  * Male or female adults (≥ 18 years) diagnosed with ITP according to the new consensus guidelines
  * No indication of a disease which may cause thrombocytopenia other than ITP.
  * Having taken eltrombopag for at least 4 months prior to beginning of study.
  * Subject experienced no toxicity other than transient eltrombopag-related toxicity or other drug intolerance.
  * Subjects treated with concomitant ITP medications (e.g. corticosteroids or azathioprine) must be receiving a dose that has been stable for at least four weeks prior to start of this study.
  * A subject is practicing an acceptable method of contraception (documented in chart). female subjects or female partners of male subjects must either be of non-child bearing potential (hysterectomy, bilateral ovariectomy, bilateral tubal ligation or post menopausal for more than one year) OR of child bearing potential using one of the following highly effective methods of contraception.
* complete abstinence from intercourse
* Intrauterine device (IUD)
* Two forms of barrier contraception. diaphragm plus spermicide, or for males condoms plus spermicide.
* Male partner is sterile and is the only partner of the female.
* Systemic contraceptives (combined oral progesterone only)

Exclusion Criteria:

A subject is at least temporarily ineligible for the study if any of the following criteria apply:

* Any clinically relevant abnormality, other than chronic ITP, identified on the screening examination, or any other medical condition or circumstance, which in the opinion of the investigator makes the subject unsuitable for participation in the study such as:

  * an active malignancy
  * an arterial or venous thrombosis
  * development of grade III-IV cardiovascular disease (including congestive heart failure, New York Heart Association (NYHA Grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation), or subjects with a QTc >480 msec.
* Recent history of alcohol/drug abuse.
* Subjects recently treated with drugs that affect platelet function (including but not limited to aspirin, clopidogrel and/or NSAIDs) or anti-coagulants for > 3 consecutive days within 2 weeks of the study start and until the end of the study.
* development of platelet agglutination abnormality that prevents reliable measurement of platelet counts.

Rescreening is possible if the condition resulting in the failed screening has been resolved. There will be no limit on the number of screening tests and the screening will be valid for 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ITP patients discontinuing the use of eltrombopag
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-06; Primary Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Platelet Response | 6 months
  To determine the frequency of a sustained response of at least 6 months in subjects with persistent or chronic ITP who have been receiving eltrombopag for a minimum of four months and are able to discontinue it within two years of initiating the tapering

CONTACTS AND LOCATIONS:
Overall Officials: James B. Bussel, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided